CLINICAL TRIAL: NCT06648278
Title: The Patient Care Outreach, Navigation, Technology and Support 2.0 Study
Brief Title: Patient Care Outreach, Navigation, Technology and Support 2.0
Acronym: COUNTS2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 22054; NCI-2024-08188 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2024-10-16; First posted 2024-10-18 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Cardiovascular Diseases
Keywords: Health Services
MeSH Terms: conditions — Breast Neoplasms; Cardiovascular Diseases | interventions — Patient Navigation; Quality of Life; Restraint, Physical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health services research (Patient COUNTS2) (Experimental): Participants attend focus groups to help further develop the patient portal and navigation program to expand to other groups. Participants use in-person navigation program and complete data collection and surveys over 15 minutes via web portal at baseline and 6 months and user experience survey at end of program participation.
  Interventions: Behavioral: Patient Navigation Program; Other: Quality-of-Life (QOL) Assessment; Other: Survey Administration

INTERVENTIONS:
Behavioral: Patient Navigation Program — Online health tool
  Other Names: Patient Navigator Program
Other: Quality-of-Life (QOL) Assessment — Online surveys to assess QOL
  Other Names: QOL Assessment; QOL Survey
Other: Survey Administration — Ancillary studies
  Other Names: Experience Survey

SUMMARY:
This is a feasibility study employing virtual patient navigation for underserved individuals who speak English, Chinese or Spanish and were diagnosed with breast cancer or cardiovascular disease to determine the extent of usability for a virtual patient navigation portal serving people in underserved communities. While not able to entirely replace in-person interactions, virtual patient navigation may be used to expand reach and availability of navigation services to a much greater segment of the population.

DETAILED DESCRIPTION:
Patient COUNTS 2.0 aims to improve and scale up the current Patient COUNTS program.

PRIMARY OBJECTIVES:

I. Identify underserved individuals who speak English, Chinese or Spanish and were diagnosed with breast cancer or cardiovascular disease through collaboration with Zuckerberg San Francisco General Hospital (ZSFG), University of California, San Francisco clinics (Athena), University of California, San Francisco registries (via medical chart review), San Francisco State University, and other community organization collaborators.

II. Conduct outreach to potential participants to let them know about the availability of virtual patient navigation via the Patient Care Outreach, Navigation, Technology and Support (COUNTS) web portal, and the Patient COUNTS patient navigation program (NCT03867916).

III. Provide patient navigation virtually.

OUTLINE:

The patient COUNTS portal will be available in English and expanded to include content in Chinese and Spanish. An initial cohort of focus group of 15 breast cancer patients, 5 navigators, social workers, caregivers or other person involved in breast cancer care will help develop the culturally and language specific components of the COUNTS program. Following implementation, breast cancer participants and cardiovascular participants will participate in an online navigation program along with family members of the patient community will be enrolled. Participants will use the online COUNTS portal to access navigation program and may choose to have online/virtual navigation support or in-person navigation support. Participants also complete data collection and surveys over 15 minutes via web portal at baseline and 6 months and user experience survey at end of program participation.

ELIGIBILITY:
Inclusion Criteria:

For Focus groups:

* Breast cancer patients: Diagnosed with breast cancer, ages 18 or older, speaks English, Mandarin/Cantonese, or Spanish
* Navigators: any patient navigator who has provided care to underserved populations diagnosed with cancer

For Portal Implementation phase:

* Ages 18 or older
* Speaks English, Mandarin/Cantonese, Spanish,
* Has any stage breast cancer
* Has access to a phone that is able to receive text messages, is willing to stay in the study for six-seven months.

Family User experience survey:

* Family member or friend who may have assisted breast cancer participant with registration, accessing or otherwise assisting breast cancer family member or friend participant with the online portal.

Exclusion Criteria:

* Any medical or psychological conditions precluding informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2023-08-10 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who reported satisfaction with COUNTS program | Up to 6 months
  Participant satisfaction will be assessed via a response of "satisfied" or "very satisfied" to survey item on satisfaction with Patient COUNTS navigation program
Rate of Participation | Up to 6 months
  Participation is defined as having at least one contact with patient navigator
Utilization rate | Up to 6 months
  Utilization is defined as the number of interactions with the patient navigator

SECONDARY OUTCOMES:
Mean scores on the Functional Assessment of Cancer Therapy- Breast (FACT-B) | Up to 6 months
  The FACT-B is a self-report instrument that measures multidimensional quality of life (QOL) in patients with breast cancer. The FACT-B consists of 37 questions that address physical, social, emotional, and functional well-being, with specific questions relevant to women with breast cancer. Each item has a score range of 0 (Not at all) to 4 (Very much), with a total score ranging from 0-148. The higher the score, the better the QOL reported by the participant.

CONTACTS AND LOCATIONS:
Overall Officials: Scarlett L Gomez, PhD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - Zuckerberg San Francisco General Hospital, San Francisco, California
  - University of California, San Francisco, San Francisco, California

IPD SHARING:
Plan to Share IPD: No